CLINICAL TRIAL: NCT06376812
Title: No Time to Pause: Physical Activity to Improve Health and Well-being of Midlife Hispanic Women During the Menopausal Transition
Brief Title: No Time to Pause: Physical Activity to Improve Health of Midlife Hispanic Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-0320
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Elevated Blood Pressure; Perimenopause
Keywords: Physical activity; Women's health; Minority health; Behavior change; Hypertension prevention
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity intervention (Experimental): Multi-level intervention to increase physical activity
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention — Physical activity

SUMMARY:
This study will test the effects of a physical activity intervention among midlife Hispanic women.

DETAILED DESCRIPTION:
The menopausal transition in midlife is a critical juncture where women experience life transitions and adverse physiological and psychological changes that increase the risk for hypertension and cardiovascular diseases in later life. Physical activity improves blood pressure, biomarkers of hypertension, sleep, mood, and well-being; however, Hispanic women meet physical activity recommendations at lower levels than non-Hispanic White women. The investigator will examine the feasibility of the physical activity intervention among sedentary midlife Hispanic women in the menopausal transition with elevated blood pressure, exploring changes in physical activity and health.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Hispanic by self-report
3. Able to speak and read English
4. Sedentary
5. Age 45-50
6. Diagnosed with elevated blood pressure or objectively measured systolic blood pressure 120-139 mmHg and/or diastolic blood pressure 80-89 mmHg averaged from ≥ 2 measures on ≥ 2 outpatient visits
7. Symptoms consistent with the menopause transition (persistent difference of ≥7 days in the length of consecutive cycles; persistence is defined as recurrence within 10 cycles of the first variable length cycle)
8. Apparently healthy
9. Self-reported ability to engage in moderate intensity physical activity
10. Access to a smart device that is compatible with a Fitbit application

Exclusion Criteria:

1. Self-reported physical activity of ≥150 minutes per week
2. Answered yes to any question on the Physical Activity Readiness (PAR-Q+) questionnaire
3. Post-menopausal (12-months without a menstrual cycle)
4. Diagnosed hypertension
5. Cardiovascular, respiratory, neurological, renal, endocrine, gastrointestinal and/or psychiatric diseases, or any cancers
6. Previous hysterectomy, oophorectomy, and/or uterine ablation
7. Medication to treat hypertension, elevated glucose, cholesterol, depression, anxiety, and insomnia
8. Hormonal medication via any route or implants
9. Tamoxifen
10. Pregnant, planning to become pregnant, or breastfeeding
11. Planning to move out of the Galveston/Houston area in the next 18 months
12. Current participation in another physical activity study or program

Ages: 45 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2027-01-20 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Days the activity monitor was worn | Baseline to 6-months
  Objectively measured days the wearable activity monitor was worn during the intervention period

SECONDARY OUTCOMES:
Physical activity as measured by minutes of moderate-vigorous intensity physical activity at 6 months | Baseline to 6-months
  Mean daily minutes of moderate-vigorous intensity physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of moderate-vigorous intensity physical activity at 6 months | Baseline to 12-months
  Mean daily minutes of moderate-vigorous intensity physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of moderate intensity physical activity at 6 months | Baseline to 6-months
  Mean daily minutes of moderate intensity physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of moderate intensity physical activity at 6 months | Baseline to 12-months
  Mean daily minutes of moderate intensity physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of vigorous intensity physical activity at 6 months | Baseline to 6-months
  Mean daily minutes of vigorous intensity physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of vigorous intensity physical activity at 6 months | Baseline to 12-months
  Mean daily minutes of vigorous intensity physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of light intensity physical activity at 6 months | Baseline to 6-months
  Mean daily minutes of light intensity physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of light intensity physical activity at 6 months | Baseline to 12-months
  Mean daily minutes of light intensity physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of total physical activity at 6 months | Baseline to 6-months
  Mean daily minutes of total physical activity taken from accelerometers for a 7 day period
Physical activity as measured by minutes of total physical activity at 6 months | Baseline to 12-months
  Mean daily minutes of total physical activity taken from accelerometers for a 7 day period
Systolic blood pressure | Baseline to 6-months
  Change in systolic blood pressure (mmHg)
Systolic blood pressure | Baseline to 12-months
  Change in systolic blood pressure (mmHg)
Diastolic blood pressure | Baseline to 6-months
  Change in diastolic blood pressure (mmHg)
Diastolic blood pressure | Baseline to 12-months
  Change in diastolic blood pressure (mmHg)

OTHER OUTCOMES:
Abdominal circumference | Baseline to 6-months
  Change in abdominal circumference (cm)
Abdominal circumference | Baseline to 12-months
  Change in abdominal circumference (cm)
Body mass index | Baseline to 6-months
  Change in body mass index (kg/m2)
Body mass index | Baseline to 12-months
  Change in body mass index (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lorenzo, PhD, RN, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The research data from this project will be deposited with a service of the Inter-university Consortium for Political and Social Research (ICPSR), openICPSR, to ensure that the research community has long-term access to the data.
Supporting Information: Study Protocol, SAP
Time Frame: We agree to deposit and/or make available our data upon completion of the clinical trial and acceptance of the data for publication. Data will be stored in the repository for at least 3 years, as required by federal retention guidelines.
Access Criteria: Data will be shared via openICPSR as open access.